CLINICAL TRIAL: NCT05071703
Title: Evaluation of TRILACICLIB in Chinese Patients With Extensive-stage Small Cell Lung Cancer (ES-SCLC) for Chemotherapy-induced Myelosuppression, Antitumor Effects of Combination Regimens, and Safety in a Real-world Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trila-CN-RWS-001
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2021-09

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — trilaciclib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trilaciclib, carboplatin, etoposide, Topotecan (Experimental): Trilaciclib plus Carboplatin combined with Etoposide OR Topotecan (ES-SCLC patients)
  Interventions: Drug: Trilaciclib

INTERVENTIONS:
Drug: Trilaciclib — * Carboplatin combined with Etoposide (ES-SCLC patients)
  * plus Topotecan (second/third line ES-SCLC patients)
  Other Names: Trilaciclib, carboplatin, etoposide#or Topotecan

SUMMARY:
This is a single-arm, real-world study in Chinese patients with extensive stage small cell lung cancer. The purpose of this study was to evaluate Trilaciclib's protection against chemotherapy-induced bone marrow suppression, the safety and the impact on the antitumor effects of the combination with chemotherapy in Chinese patients with ES-SCLC in the real world. Patients with ES-SCLC who already use or plan to use Trilaciclib will be invited to participate in the study. Data were collected from 28 days prior to initial chemotherapy (platinum/etoposide or topotecan systemic chemotherapy) after patients signed informed consent until patients died, dropped out of the study, lost to follow-up, informed withdrawal, or study termination. The end time of the study was defined as withdrawal of information, loss of follow-up or death of all enrolled patients, or 12 months after the last patient was enrolled, whichever happened earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign informed consent;
2. must be at least 18 years when fisrt dose of Trilaciclib, regardless of gender:
3. Patients with extensive small-cell lung cancer confirmed by histology or cytology
4. Patients suitable for Trilaciclib combined with platinum/etoposide or Trilaciclib combined with topotecan treatment

Exclusion Criteria:

1. Patient is currently participating in other Interventional clinical studies;
2. Patients received systemic chemotherapy other than the regimens recommended in inclusion criteria 4 During Trilaciclib treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of severe neutropenia (SN) | during Trilaciclib plus chemotherapy assessed up to 6 months
  Incidence of severe neutropenia (SN)

SECONDARY OUTCOMES:
Incidence of grade 3 and 4 hematologic toxicity | during Trilaciclib plus chemotherapy assessed up to 6 months
Incidence of intravenous or oral antibiotic administration in treatment | during Trilaciclib plus chemotherapy assessed up to 6 months
Incidence of G-CSF treatment | during Trilaciclib plus chemotherapy assessed up to 6 months
Changes of absolute neutrophil count, platelet count, absolute lymphocyte count (ALC) and hemoglobin over time | during Trilaciclib plus chemotherapy assessed up to 6 months
Incidence of red blood cell (RBC) transfusions at or after week 5 | during Trilaciclib plus chemotherapy assessed up to 6 months
The incidence of ESA administration in treatment | during Trilaciclib plus chemotherapy assessed up to 6 months
The incidence of TPO administration in treatment | during Trilaciclib plus chemotherapy assessed up to 6 months
The incidence of platelet transfusion | during Trilaciclib plus chemotherapy assessed up to 6 months
The number and frequency of all-caused chemotherapy drugs reduction | during Trilaciclib plus chemotherapy assessed up to 6 months
composite end point - Significant hematologic adverse event (occurrence of any of the following events：all-cause hospitalization; all-cause dose reduction; Febrile neutropenia; Severe neutropenia ) | during Trilaciclib plus chemotherapy assessed up to 6 months
Incidence of infectious serious adverse events | during Trilaciclib plus chemotherapy assessed up to 6 months
Incidence of pulmonary infection serious adverse events | during Trilaciclib plus chemotherapy assessed up to 6 months
The incidence of febrile neutropenia | during Trilaciclib plus chemotherapy assessed up to 6 months
Objective response rate | during Trilaciclib plus chemotherapy assessed up to 6 months
duration of response | during Trilaciclib plus chemotherapy assessed up to 6 months
Progression-free survival time | during Trilaciclib plus chemotherapy assessed up to 6 months
Disease control rate | during chemotherapy assessed up to 6 months
verall survival | maximun up to 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yongxing Chen, Principal Investigator — Hainan General Hospital
Locations (1):
- Hainan General Hospital, Haikou, Hainan, China